CLINICAL TRIAL: NCT04166331
Title: Adjunctive DobutAmine in sePtic Cardiomyopathy With Tissue Hypoperfusion: a Randomized Controlled Multi-center Trial
Brief Title: Adjunctive DobutAmine in sePtic Cardiomyopathy With Tissue Hypoperfusion
Acronym: ADAPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Centre d'Investigation Clinique 1415 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 87RI18_0012 (ADAPT)
Record Dates: First submitted 2019-10-25; First posted 2019-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Cardiomyopathies; Hypoperfusion; Left Ventricular Systolic Dysfunction
Keywords: sepsis; Cardiomyopathies; Hypoperfusion; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Sepsis; Cardiomyopathies; Ventricular Dysfunction, Left | interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Placebo will initially be started at a dose of 2.5 µg/kg/min and subsequently titrated using incremental steps (predefined durations) of 2.5 µg/kg/min, up to a maximal dose of 10 µg/kg/min
  Interventions: Drug: Placebos
- Experimental (Experimental): Dobutamine will initially be started at a dose of 2.5 µg/kg/min and subsequently titrated using incremental steps (predefined durations) of 2.5 µg/kg/min, up to a maximal dose of 10 µg/kg/min
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Placebos — Placebo will initially be started at a dose of 2.5 µg/kg/min and subsequently titrated using incremental steps (predefined durations) of 2.5 µg/kg/min, up to a maximal dose of 10 µg/kg/min. Dose adaptation will be left at the discretion of attending physician.
  Arms: Control
Drug: Dobutamine — Dobutamine will initially be started at a dose of 2.5 µg/kg/min and subsequently titrated using incremental steps (predefined durations) of 2.5 µg/kg/min, up to a maximal dose of 10 µg/kg/min. Dose adaptation will be left at the discretion of attending physician.
  Arms: Experimental

SUMMARY:
Sepsis induces both a systolic and diastolic cardiac dysfunction. The prevalence of this septic cardiomyopathy ranges between 30 and 60% according to the timing of assessment and definition used. Although the prognostic role of septic cardiomyopathy remains debated, sepsis-induced left ventricular (LV) systolic dysfunction may be severe and associated with tissue hypoperfusion, while it appears to fully recover in survivors. Accordingly, optimization of therapeutic management of septic cardiomyopathy may contribute to improve tissue hypoperfusion in increasing oxygen delivery, and to reduce related organ dysfunctions in septic shock patients.

Echocardiography is currently the recommended first-line modality to assess patients with acute circulatory failure.

Current Surviving Sepsis Campaign strongly recommends Norepinephrine as the first-choice vasopressor in fluid-filled patients with septic shock. In contrast, the use of Dobutamine is only suggested (weak recommendation, low quality of evidence) in patients with persistent tissue hypoperfusion despite adequate fluid resuscitation and vasopressor support. Levosimendan, an alternative inodilator, has failed preventing acute organ dysfunction in septic patients and has induced more supraventricular tachyarrhythmias than in the control group. Data supporting Dobutamine in this setting are scarce and primarily physiologic and based on monitored effects of this drug on hemodynamics and indices of tissue perfusion.

No randomized controlled trials have yet compared the effects of Dobutamine versus placebo on clinical outcomes. In open-labelled, small sample trials, the ability of septic patients to increase their oxygen delivery during Dobutamine administration appears to be associated with lower mortality.

The tested hypothesis in the ADAPT trial is that Dobutamine will reduce tissue hypoperfusion and associated organ dysfunctions in patients with septic shock and associated septic cardiomyopathy. In doing so, it may participate in improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years hospitalized in ICU
* > Septic shock (Sepsis-3 definition):

  1. Clinically suspected or documented acute infection
  2. Responsible for organ dysfunction(s): change in SOFA ≥ 2 points
  3. With persisting hypotension (systolic and/or mean arterial pressure < 90 / < 65 mmHg) despite adequate fluid resuscitation (≥ 30 mL/kg, unless presence of pulmonary venous congestion)
  4. Requiring vasopressor support (Norepinephrine) to maintain steady mean arterial pressure ≥ 65 mmHg
  5. And lactate > 2 mmol/L
* Septic cardiomyopathy: echocardiographically measured LV ejection fraction (EF) ≤ 40% and LV outflow tract velocity-time integral < 14 cm
* Informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Hypersensitivity to Dobutamine, 5% Dextrose, or to the excipients
* Ventricular rate > 130 bpm (sinus rhythm or not)
* Severe ventricular arrhythmia
* Obstructive cardiomyopathy with pressure gradient at rest ≥ 50 mmHg unrelated to uncorrected hypovolemia
* Severe aortic stenosis: mean gradient > 40 mmHg, peak aortic jet velocity > 4 m/s, aortic valve area < 1 cm² (aortic valve area index < 0.6 cm²/m²)
* Acute coronary syndrome
* Decision to limit care or moribund status (life expectancy < 24 h)
* Absence of affiliation to Social Security
* Subjects under juridical protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score evolution | Day 0 to Day 3
  Evolution of a modified Sequential (Sepsis-Related) Organ Failure Assessment (SOFA) score (no gradation of the neurologic system) between baseline (before randomization) and Day 1, Day 2 and Day 3 after randomization. Min value =0. Max value =20 . The highest score means the worst situation

SECONDARY OUTCOMES:
Circulating lactate level measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Biological indices of tissue dysoxia at baseline, hour 6, Day1, Day 2 and Day 3 after initiating Dobutamine / placebo
Central venous oxygen saturation (ScvO2) measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Biological indices of tissue dysoxia at baseline, hour 6, Day1, Day 2 and Day 3 after initiating Dobutamine / placebo
Open-labelled Dobutamine dayly maximal dose used as rescue therapy | through study completion, an average 90 days
  Requirement of organ function supports during ICU stay. Maximal dose in mcg/kg/min of open-labelled Dobutamine used as rescue therapy
Open-labelled Dobutamine duration used as rescue therapy | through study completion, an average of 90 days
  Requirement of organ function supports during ICU stay. Duration in days of open-labelled Dobutamine used as rescue therapy
Vasopressor support duration | through study completion, an average of 90 days
  Requirement of organ function supports during ICU stay. Duration in days of vasopressor support
Vasopressor support dayly maximal dose | through study completion, an average of 90 days
  Requirement of organ function supports during ICU stay. Maximal dose in mg/h by day of vasopressor support
Invasive mechanical ventilation duration | through study completion, an average of 90 days
  Requirement of organ function supports during ICU stay. Duration of invasive mechanical ventilation
Renal replacement therapy number | through study completion, an average of 90 days
  Requirement of organ function supports during ICU stay. Number of session of renal replacement therapy (excluding hemodialysis patient for chronic renal failure at the time of randomization)
Renal replacement therapy duration | through study completion, an average of 90 days
  Requirement of organ function supports during ICU stay. Duration of renal replacement therapy (excluding hemodialysis patient for chronic renal failure at the time of randomization)
Arterial pressure measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Systolic, diastolic and mean arterial blood pressure (in mmHg) at Baseline, h6, Day 1, Day 2 and Day3after initiating Dobutamine / placebo
heart rate measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Heart rate measurement in bpm at Baseline, Hour 6, Day 1, Day 2 and Day3 after initiating Dobutamine / placebo
Central venous pressure measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Central venous pressure in cm H2O at Baseline, Hour 6, Day 1, Day 2 and Day3 after initiating Dobutamine / placebo
Cardiac index measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Cardiac index measurement in L/min/m2 at Baseline, Hour 6, Day 1, Day 2 and Day3 after initiating Dobutamine / placebo
Stroke volume measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Stroke volume measurement in mL status at Baseline, Hour 6, Day 1, Day 2 and Day3 after initiating Dobutamine / placebo
Hypotension measurement | Hour 0, Hour 6, Day 1, Day 2 and Day 3
  Severe cardiovascular adverse events from inform consent to ICU discharge : Hypotension related to worsened vasoplegia
Supraventricular arrhythmias measurement | through study completion, an average of 90 days
  Severe cardiovascular adverse events from inform consent to ICU discharge. Supraventricular arrhythmias with ventricular rate > 140 bpm
Ventricular arrhythmias measurement | through study completion, an average of 90 days
  Severe cardiovascular adverse events from inform consent to ICU discharge. Ventricular arrhythmias
Occurence of Acute coronary syndrome | through study completion, an average of 90 days
  Severe cardiovascular adverse events from inform consent to ICU discharge. Acute coronary syndrome
Occurence of Stroke | through study completion, an average of 90 days
  Severe cardiovascular adverse events during ICU stay. Stroke
Mortality | Day 90
  Number of death
Mortality causes | Day 90
  Cause of death
Organ function free supports | Day 90
  Number of days free from vasopressor support, invasive mechanical ventilation, renal replacement therapy from inform consent to ICU discharge
Number of days in ICU and hospital | Day 90
  Length of ICU and hospital stay
echocardiographic assessment of left ventricular systolic function | Day 0 and Day 1
  ejection fraction measurement
Leucocyte subsets level | Hour 6
  Leucocyte subsets level according to the severity of the sepsis-induced LV systolic dysfunction and hemodynamic effects of the study drug administration
Cytokines level | Hour 6
  tumor necrosis factor (TNF) -α, Interferon ɣ, Interleukin-6, 8 and 10 cytokines concentration will be assess according to the severity of the sepsis-induced LV systolic dysfunction and hemodynamic effects of the study drug administration. Result for each cytokine concentration will be given in picograms per milliliter.
LV global longitudinal strain measurement | Hour 6, Day 1, Day 2 AND Day 3
  LV segmental deformation longitudinal analysis
RV free wall strain measurement | Hour 6, Day 1, Day 2 AND Day 3
  deformation of right ventricular myocardial tissue / routinely using with echocardiography or post exam analysis
LV volume measurement | Hour 6, Day 1, Day 2 AND Day 3
  Ratio between systolic and diastolic left ventricular volume / routinely using with echocardiography
LV ejection fraction measurement | Hour 6, Day 1, Day 2 AND Day 3
  Cardiac output measurement with echocardiography Doppler (in centers routinely using transpulmonary thermodilution). Quality of left ventricular contraction
RV volume measurement | Hour 6, Day 1, Day 2 AND Day 3
  Ratio between systolic and diastolic right ventricular volume / routinely using with echocardiography
RV ejection fraction measurement | Hour 6, Day 1, Day 2 AND Day 3
  Cardiac output measurement with echocardiography Doppler (in centers routinely using transpulmonary thermodilution). Quality of right ventricular contraction
Transpulmonary thermodilution measurement | Hour 6, Day 1, Day 2 AND Day 3
  In selected centers routinely using continuous monitoring of cardiac output using transpulmonary thermodilution: agreement of cardiac output measurement with echocardiography Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: VIGNON Philippe, MD, Principal Investigator — University Hospital, Limoges
Locations (21):
- France (21):
  - CHU Orléans - service de Réanimation, Orléans, Orleans
  - CHU Strasbourg - service de Réanimation, Strasbourg, Strasbourg
  - CHU Tours - Service de Réanimation, Tours, Tours
  - Angouleme Hospital, Angoulême
  - Argenteuil Hospital, Argenteuil
  - CH de Bethune, Béthune
  - University Hospital, Brest
  - CH de Brive, Brive-la-Gaillarde
  - CH de Cannes, Cannes
  - Aphp - Henri Mondor, Créteil
  - Dijon university hospital, Dijon
  - CH d'Haguenau, Haguenau
  - Le Mans Hospital, Le Mans
  - Lille University Hospital, Lille
  - Limoges University Hospital, Limoges
  - HCL, Lyon
  - Montpellier University Hospital, Montpellier
  - Nice University Hospital, Nice
  - Aphp - Ambroise Paré, Paris
  - Poitiers University Hospital, Poitiers
  - CH de Toulon, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vignon P, Leger J, Evrard B, Goudelin M, Vaidie J, Brit S, Giraudeau B. Adjunctive dobutamine in patients with septic cardiomyopathy and tissue hypoperfusion: a blinded randomised controlled multicentre trial study protocol of the ADAPT-dobutamine trial. BMJ Open. 2025 Jun 30;15(6):e101200. doi: 10.1136/bmjopen-2025-101200. PMID 40588393